CLINICAL TRIAL: NCT06141616
Title: Effects of Pulmonary Rehabilitation on Activities of Daily Living, Physical Activities of Daily Living and Other Clinical Outcomes in Children With Asthma: a Randomized Clinical Trial
Brief Title: Effects of Pulmonary Rehabilitation on Clinical Outcomes in Children With Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Karina Furlanetto, Professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PuzziVC_PhD_FurlanettoKC
Record Dates: First submitted 2023-11-11; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Asthma in Children; Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Sessions once a week, covering information about the pathophysiology of asthma, medication instructions, self-monitoring techniques, environmental control techniques, and prevention strategies for children, adolescents, and families. They will also receive physical activity recommendations, as well as information about the importance and benefits of being physically active and maintaining a healthy lifestyle. The sessions will feature educational and playful videos, presentations, and participants will be able to clarify their doubts about the topic addressed.
  Interventions: Other: Asthma Rehabilitation Program
- Experimental group (Experimental): Rehabilitation program performed 3x/week. Each session will last 60 minutes, with a minimum interval of 24 hours, for a period of three months. The main focus of the intervention is aerobic training, which will be carried out in three stages, treadmill with a warm-up (10 minutes), load (20 minutes), and cool-down (5 minutes). With an initial intensity of 65% of the maximum load obtained in the incremental shuttle walk test (ISWT). The intensity will be gradually increased up to 115%, keeping dyspnea and fatigue values between 4 and 6, according to the modified Borg scale. In addition, we will do a circuit focused on aerobic activities, maintaining target heart rate during its performance for 20 minutes. When necessary, supplemental oxygen will be provided during training. Volunteers in this group will receive a bronchodilator dose before starting each day's session. This group will hold educational sessions as well.
  Interventions: Other: Asthma Rehabilitation Program

INTERVENTIONS:
Other: Asthma Rehabilitation Program — The group will receive free physiotherapy treatment with aerobic exercises, 3x/week, 60 minutes a day, lasting 3 months, in addition to educational sessions in a playful way.

SUMMARY:
Although the practice of physical activity is recommended for children with asthma, the scientific literature available so far has focused mainly on improving functional capacity and quality of life. However, the effects of pulmonary rehabilitation in this population, especially in improving the level of physical activity in daily living (PADL) and activities of daily living (ADLs) have not yet been investigated in depth. Therefore, the objective of this study is to verify the effects of pulmonary rehabilitation on PADL, ADL, and other clinical outcomes of children with asthma. For this, a randomized clinical trial will be carried out that will have 2 groups: the control group (CG), which will receive only educational sessions, and the intervention group (IG) which will participate in a pulmonary rehabilitation program with supervised aerobic training performed three times a week with sessions of 60 minutes each. The total duration of interventions in both groups will be 12 weeks. The primary outcomes of this study are PADL (assessed using a physical activity monitor - Actigraph) and ADL; however, the following will also be evaluated: lung function, functional capacity, asthma control, and quality of life. We hypothesized that the performance of regular physical activity and supervised physical exercise by individuals with asthma could positively impact health outcomes with better control of asthma symptoms, better performance in ADL and PADL, and better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 12 years old;
* Clinical diagnosis of asthma, established according to the criteria of the Global Initiative for Asthma (GINA);
* Absence of other lung diseases or signs and symptoms of other lung diseases;
* Absence of cognitive changes;
* Absence of signs and symptoms of gastroesophageal reflux disease and dysphagia;
* Clinical stability according to the criteria of the Global Initiative for Asthma (GINA);

Exclusion Criteria:

* Desire of the patient and/or the patient's family to discontinue participation in the study for any reason;
* Present some new limitations that may interfere with functionality;
* Comorbidities that prevent or contraindicate the performance of the proposed interventions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 12 weeks from randomization
  Number of steps per day, time spent (in minutes and percentage of the day) in light-intensity and moderate to vigorous physical activities, measured by a triaxial activity monitor.
Sedentary behavior | 12 weeks from randomization
  Time spent (in minutes and percentage of the day) in sedentary activities, measured by a triaxial activity monitor.
The activity of daily living | 12 weeks from randomization
  Time on a specific test to evaluate activities of daily living in children

SECONDARY OUTCOMES:
Initial assessment about general characteristics and health status | 12 weeks from randomization
  A questionnaire will be prepared to cover all these topics: age, weight, height, body mass index (BMI), history of prematurity, personal, family, and surgical history, in addition to comorbidities. These data will be used to characterize the sample and the questionnaire will be answered with the help of the family member.
Pulmonary Function | 12 weeks from randomization
  Spirometry determining the forced expiratory volume in the first second (FEV1), forced vital capacity (FVC) and FEV1/ FVC index.
Asthma Control | 12 weeks from randomization
  The asthma control questionnaire (ACT or ACT-C) will be applied according to the child's age, to determine if the asthma is controlled. The ACT consists of five questions. The score for each question varies between 1 and 5 points. The minimum score of the questionnaire is 5 points and the maximum score is 25 points. The ACT-C, which will be applied to children younger than 11 years and 12 months, consists of seven questions, four of them answered by the child and three by parents or guardians, with a minimum score of 0 and a maximum of 27.
Exacerbation and medication diary | 12 weeks from randomization
  Diaries will be given to patients in which individuals with asthma or their guardians must record any asthma exacerbations, as well as the use of medications for the disease. Exacerbations will be defined as the use of oral corticosteroids due to worsening symptoms; the need for a doctor's appointment or emergency care due to worsening symptoms. These data may be used as confounding factors in the statistical analysis in case of eventual exacerbations and/or changes in medications during the intervention.
Quality of life in asthma | 12 weeks from randomization
  The Pediatric Asthma Quality Of Life Questionnaire (PAQLq), consists of 23 questions divided into three domains: physical activity limitations, symptoms, and emotions. Responses will be measured on a 7-point scale, where 1 indicates maximum loss and 7 indicates no loss. This questionnaire has already been translated and validated for the Brazilian language, for the population of children and adolescents with asthma and the other questionnaire used to assess quality of life in children, the Pediatric Quality of Life (PedsQL), Structurally, it consists of 27 items divided into 8 subscales: pain and injuries, nausea, anxiety about the procedure, anxiety about the treatment, concerns, difficulties cognitive, perception of physical appearance, communication. The scale consists of 5 response options, like "Likert": "never", "rarely", "sometimes", "often", and "almost always" .
Sleep assessment | 12 weeks from randomization
  Children's Sleep Habits Questionnaire (CSHQ) assesses parents' perception of their children's sleep during the previous week or, if not representative for some reason, during a more recent typical week. The frequency of sleep behaviors is rated on a three-point scale, such as "usually" (five to seven times a week, totaling three points), "sometimes" (two to four times a week, totaling two points), or " rarely" (0 to once a week, totaling one point).
Parents' knowledge about the child's illness | 12 weeks from randomization
  Asthma Knowledge Questionnaire - Short form (AKQ) The scale contains 10 statements, and responses are given on a 5-point Likert scale, with responses ranging from "totally disagree" to "totally agree", ranging from 1 to 5 respectively. Negative items will be reverse-coded by subtracting the response value from 5. This implies that the correct answer is always "strongly agree" for all questions. The final score is the sum of all responses, ranging from 10 to 50, with higher scores indicating greater knowledge of asthma.
Family Health Questionnaire | 12 weeks from randomization
  The purpose of this questionnaire is to obtain information about the health behavior of those responsible and the health behavior of the child. Answering the questionnaire will take about 45 minutes of the parents' time and will be applied while the child performs the functional tests.
Report of performance in physical activities | 12 weeks from randomization
  Preschool-age Children's Physical Activity Questionnaire (Pre-PAQ) and Physical Activity Questionnaire for Children (PAQ-C) according to age.
Motivation scale | 12 weeks from randomization
  A simple question based on the transtheoretical model of behavior change about self-reported motivation and physical activity behavior will be applied to children.
Submaximal exercise capacity | 12 weeks from randomization
  To assess this outcome, the six-minute walk test (6MWT) and sit-to-stand (STS) will be used. The 6MWT will be performed according to international standards. Individuals will be instructed to cover the longest possible distance in 6 minutes in a 30-meter-long flat corridor, without running. Two tests will be performed with a minimum interval of 30 minutes. Sit-to-stand: The test will be performed using a chair that ensures 90 degrees of hip, knee, and ankle flexion. When individuals are instructed with the word "go", they will have to get up immediately without delay and sit down again, repeating the procedure as many times as they can within 1 minute, the number of repetitions will be counted.
Maximal exercise capacity | 12 weeks from randomization
  Incremental Shuttle Walk Test (ISWT): The ISWT will be performed in a 10 m-long corridor as per the original description. It is a test externally cadenced by a sound signal, in which the speed increases every minute, ranging from 1.79 to 10.2 km/h. The total test time and the distance covered by the patient will be recorded at the end of the test

CONTACTS AND LOCATIONS:
Overall Officials: Vitória Puzzi, Msc, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Centro de Pesquisa e Pós Graduação na Unopar, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No